CLINICAL TRIAL: NCT06559761
Title: Image Driven Hepatocellular Carcinoma Invasiveness Evaluation Research
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Other Study IDs: S2024-423
Record Dates: First submitted 2024-08-06; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma Stage III
Keywords: Hepatocellular Carcinoma; Prognosis; Imaging; Gross classification
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Resected tumor specimen will be used for histological assessment and DNA/mRNA sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TYPE I: Gross classification of resected specimen: single nodule with distinct margin, usually round with complete tumour envelope
  Interventions: Procedure: Hepatectomy
- TYPE II: Gross classification of resected specimen: single nodule with extranodular growth, no more than three extranodular points
  Interventions: Procedure: Hepatectomy
- TYPE III: Gross classification of resected specimen: a unifocal lesion composed of confluent multiple nodules, distinct boundaries among the nodules
  Interventions: Procedure: Hepatectomy
- TYPE IV: Gross classification of resected specimen: infiltrative nodule, with poor demarcated boundary and especially multiple extranodular points
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — According to guideline recommended procedure of hepatectomy

SUMMARY:
Hepatocellular carcinoma (HCC) is a highly heterogeneous malignant tumor with significant differences in invasion, proliferation ability and patient prognosis. Currently, there is a lack of non-invasive and simple indicators to predict the prognosis of HCC patients and assist clinical decision-making. The identification of HCC macroscopic or histopathological classification requires large pathological specimens obtained through surgical resection, but only about 20% of patients are eligible for surgical treatment. Moreover, most liver cancer diagnoses can be confirmed by imaging examinations without relying on pathological results. For patients who have not undergone surgical resection, the lack of histopathological information during treatment means that there is no basis for judging tumor proliferation and obtaining rich prognostic information. Therefore, evaluating the invasion and proliferation ability of HCC based on macroscopic imaging assessment has important implications for guiding individualized diagnosis and treatment throughout the entire process including surgical strategy guidance, local treatment selection, systemic therapy planning as well as patient follow-up and prognosis evaluation.

Ultrasound and MRI are ideal entry points as first-line imaging methods for liver cancer diagnosis. This study aims to evaluate HCC macroscopic or histopathological classification based on multimodal imaging (ultrasound, CT, MRI), thereby assessing its invasion and proliferation ability which has important implications for guiding individualized diagnosis and treatment throughout the entire process including surgical strategy guidance, local treatment selection, systemic therapy planning as well as patient follow-up and prognosis evaluation.

By analyzing macroscopic image features we aim to explore their cross-scale correlations with HCC macroscopic classification,histopathological classification,and gene molecular typing.

ELIGIBILITY:
Inclusion Criteria:

* According to the WHO classification, the pathological diagnosis is hepatocellular carcinoma.
* The initial treatment is curative-intent hepatectomy.
* There is no evidence of major vascular/hepatic portal invasion, extrahepatic/lymph node metastasis, or other malignant tumors.
* Age 18-80 years old.

Exclusion Criteria:

· Not meeting any one of the inclusion criteria or being unwilling/unable to follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients pathologically diagnosed with hepatocellular carcinoma and underwent curative-intent hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | through study completion, an average of 1 year
  OS was defined as death related to any cause and was indexed from the date of ablation or surgery until last contact or death

SECONDARY OUTCOMES:
Disease-free survival | through study completion, an average of 1 year
  DFS was defined as the time interval between first treatment and recurrence or death, whichever occurred earlier
Imaging features | through study completion, an average of 1 year
  MRI or ultrasound Imaging features of the four types
Quantification of immune cells of the resected liver tumour | through study completion, an average of 1 year
  Quantification of immune cells of the resected liver tumour using HE staining and immunohistological staining to assess molecular marker and cell infiltration in tumor and liver parenchyma
mRNA sequencing data of the resected liver tumour and peritumor parenchyma | through study completion, an average of 1 year
  mRNA sequencing data of the resected liver tumour and peritumor parenchyma specimen to assess the gene enrichment

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided